CLINICAL TRIAL: NCT00093977
Title: An Open-label, Single-Arm Study to Assess the Safety of Darbepoetin Alfa Manufactured by a Serum Free Bioreactor Technology in Subjects With Chronic Kidney Disease
Brief Title: Study to Assess Darbepoetin Alfa in Subjects With Chronic Kidney Disease
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Amgen (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 20040180
Record Dates: First submitted 2004-10-07; First posted 2004-10-11 (Estimated); Last update posted 2013-05-24 (Estimated); Status verified 2013-05

CONDITIONS: Kidney Disease; Chronic Kidney Disease
Keywords: Chronic Kidney Disease; Dialysis; Anemia; Nephrology
MeSH Terms: conditions — Kidney Diseases; Renal Insufficiency, Chronic; Anemia

ARMS (1):
- darbepoetin alfa SF (Experimental)
  Interventions: Drug: darbepoetin alfa SF

INTERVENTIONS:
Drug: darbepoetin alfa SF — Frequency of dosing depends on frequency at randomization:
  rHuEPO QW = darbepoetin alfa SF Q2W (dosing conversion table in protocol) rHuEPO biw or tiw = darbepoetin alfa SF QW (dosing conversion table in protocol) darbepoetin alfa RB = darbepoetin alfa SF at same dose and frequency PFS 10, 15, 20, 30, 40, 50, 60, 80, 100, 150, 200 or 300 mcg; Hb maintained between 11.0 - 13.0 g/dL

SUMMARY:
The purpose of this study is to determine whether darbepoetin alfa manufactured by the current "roller bottle" technology and darbepoetin alfa manufactured by a serum free process have a comparable safety profile.

ELIGIBILITY:
Inclusion Criteria:

* Currently diagnosed with Chronic Kidney Disease, either receiving or not receiving dialysis
* Anemic
* Currently on erythropoietic therapy
* Controlled hypertension
* Clinically stable

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1100 (Estimated)
Dates: Start 2004-10; Primary Completion 2007-01 (Actual); Study Completion 2007-01 (Actual)

PRIMARY OUTCOMES:
To determine whether darbepoetin alfa manufactured by a roler bottle technology (darbepoetin alfa RB) and darbepoetin alfa manufactured by a serum free process (darbepoetin alfa SF) have a comparable safety profile | Entire Study

SECONDARY OUTCOMES:
To characterize laboratory parameters in subjects with CKD | Entire Study

CONTACTS AND LOCATIONS:
Overall Officials: MD, Study Director — Amgen

REFERENCES:
- [Result] Horowitz J, Agarwal A, Huang F, Gitlin M, Gandra SR, Cangialose CB. Empirical methods to calculate an erythropoiesis-stimulating agent dose conversion ratio in nondialyzed patients with chronic kidney disease. J Manag Care Pharm. 2009 Nov-Dec;15(9):741-50. doi: 10.18553/jmcp.2009.15.9.741. PMID 19954265
- See also: AmgenTrials clinical trials website — http://www.amgentrials.com
- See also: Notice regarding posted summaries of trial results — http://download.veritasmedicine.com/REGFILES/amgen/Amgen_results_disclaimer.pdf
- See also: To access clinical trial results information click on this link — http://download.veritasmedicine.com/REGFILES/amgen/08D_FDAMA_113_Posting_Summary_33_NESP_20040180.pdf
- See also: FDA-approved Drug Labeling — http://www.aranesp.com